CLINICAL TRIAL: NCT00478101
Title: Opioid Rotation Versus Combination for Chronic Uncontrolled Cancer Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GMO-SC-61
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Advanced Solid Cancers
Keywords: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: oxycodone fentanyl

SUMMARY:
For cancer patients with inadequate pain relief, a switch to an alternative opioid is the preferred option for symptomatic improvement. However, multiple opioids are often simultaneously administered for anecdotal reasons.

The present study isdesigned to assess the analgesic profiles of two different strategies in chronic cancer pain: the opioid rotation from oxycodone to transdermal fentanyl and the combination of oral oxycodone and transdermal fentanyl.

DETAILED DESCRIPTION:
Patients with uncontrolled cancer pain despite treatment of oral morphine equivalent ≥100 mg/d will be randomly assigned to oral opioids to transdermal fentanyl (rotation group) or oral oxycodone plus fentanyl (combination group). Patients answer a questionnaire that included pain severity (0 to 10) and interference items at baseline and after one week. Primary outcomes are change in pain score and treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Uncontrolled Pain That Required Stronger Opioid Therapy Than They Have Been Taking
* Histologically Confirmed Solid Cancer
* Aged Over 18 Years
* Admitted in a Palliative Cancer Care Unit

Exclusion Criteria:

* Uspected to Have Narcotic Abuse, Clinically Relevant CO2 Retention or Had an Active Skin Disease
* Inability to swallow oral medication, and impaired sensory or cognitive function
* Patients who had an active infection, uncontrolled central nervous system involvement, or on antitumor therapy of any kind

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2006 (Actual)
Dates: Start 2006-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change in pain score and treatment success

SECONDARY OUTCOMES:
Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Se Hoon Park, MD, Principal Investigator — Gachon University Gil Medical Center, Incheon, Korea

REFERENCES:
- [Derived] Kim HJ, Kim YS, Park SH. Opioid rotation versus combination for cancer patients with chronic uncontrolled pain: a randomized study. BMC Palliat Care. 2015 Sep 16;14:41. doi: 10.1186/s12904-015-0038-7. PMID 26377913